CLINICAL TRIAL: NCT00593905
Title: Pharmacogenomics in Pulmonary Arterial Hypertension: A Multi-Center International Study to Determine Whether in PAH Patients Clinical Associations Exist Between the Efficacy and Toxicity of Endothelin Receptor Antagonists and Several Gene Polymorphisms in Several Key Disease-Specific and Therapy Specific Genes
Brief Title: Pharmacogenomics in Pulmonary Arterial Hypertension
Status: Withdrawn | Type: Observational
Why Stopped: study not started not an ACT
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Baylor College of Medicine (Other); Emory University (Other); University of Chicago (Other); Johns Hopkins University (Other); Tufts Medical Center (Other); Sir Mortimer B. Davis - Jewish General Hospital (Other); London Health Sciences Centre (Other); University of Maryland, College Park (Other); University of California, San Francisco (Other); University of Calgary (Other); Chest Medical Associates (Unknown); Columbia University (Other); Lung Diagnostics, Ltd. (Unknown); Duke University (Other); University of California, Los Angeles (Other); Latter Day Saints Hospital (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Massachusetts General Hospital (Other); Mayo Clinic (Other); Medical College of Wisconsin (Other); Southeastern Lung Care (Unknown); Suncoast Lung Center (Unknown); Children's Hospital Colorado (Other); University Hospitals Cleveland Medical Center (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pittsburgh Medical Center (Other); University of Southern California (Other); The University of Texas Medical Branch, Galveston (Other); Vanderbilt University (Other); Wayne State University (Other); Ohio State University (Other); University of Alabama at Birmingham (Other); Washington University School of Medicine (Other); Sentara Norfolk General Hospital (Other); University of Texas Southwestern Medical Center (Other); Bay Area Chest Physicians (Other)
Responsible Party: Principal Investigator, Dawnmarie DeFazio, Professor of Medicine, Drexel University College of Medicine, James Magovern Chair for Cardiovascular Research Director and Section Head Advanced Heart Failure, Transplant, Mechanical Circulatory Support and Pulmonary Hypertension Programs, West Penn Allegheny Health System
Other Study IDs: RC-4590; RC #4590 (Other: Allegheny General Hospital)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension; PAH WHO Group I
Keywords: Pulmonary Arterial Hypertension; Pulmonary Hypertension; Pharmacogenomics; DNA Testing; sitaxsentan; bosentan; ambrisentan; elevated pulmonary artery pressures; Letairis; Tracleer; Thelin; Primary Pulmonary Hypertension; Pulmonary Artery
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension | interventions — sitaxsentan; Bosentan; ambrisentan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: GROUP 1
  1. Patients have to be currently enrolled or previously enrolled in STRIDE FPH01, FPH01-XC FPH02, FPH02x, FPH03, FPH04 or FPH06.
  2. WHO Group 1 Pulmonary arterial Hypertension: Idiopathic, Familial, Associated with (APAH) Collagen vascular disease, congenital systemic-to-pulmonary shunts, portal hypertension, Drugs and toxins (e.g., anorexigens, rapeseed oil, L-tryptophan, methamphetamine, and cocaine), other (thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders, splenectomy) Associated with significant venous or capillary involvement, Pulmonary veno-occlusive disease, Pulmonary-capillary hemangiomatosis.
  Interventions: Drug: Sitaxsentan
- Group 2: Group 2
  1. Patients currently receiving bosentan or ambrisentan OR who have previously received bosentan or ambrisentan for greater than 4 (four) months.
  2. WHO Group 1 Pulmonary Arterial Hypertension: Idiopathic, Familial, Associated with (APAH), collagen vascular disease, congenital systemic-to-pulmonary shunts, portal hypertension, drugs and toxins (e.g., anorexigens, rapeseed oil, L-tryptophan, methamphetamine, and cocaine), other (thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders, or splenectomy), associated with significant venous or capillary involvement, pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis.
  Interventions: Drug: Bosentan, Ambrisentan

INTERVENTIONS:
Drug: Sitaxsentan — Sitaxsentan sodium 100 mg tablet every morning
  Other Names: Sitaxsentan-Thelin
  Groups: Group 1
Drug: Bosentan, Ambrisentan — Bosentan 125 mg tablet twice daily Ambrisentan 5-10 mg tablet once daily
  Other Names: Bosentan-Tracleer; Ambrisentan-Letairis
  Groups: Group 2

SUMMARY:
Our goal is to determine clinically in Pulmonary Arterial Hypertension patients if associations exist between the efficacy and toxicity of sitaxsentan, bosentan, and ambrisentan and several gene polymorphisms in several key disease-specific and therapy specific genes. Also characterized is the relationship between these polymorphisms and the severity of Pulmonary Arterial Hypertension using either baseline hemodynamic or clinical surrogates for disease severity.

Hypothesis: Polymorphisms influence the efficacy and toxicity of specific Pulmonary Arterial Hypertension therapy as well as development/severity of PAH via their effect on PA remodeling, drug response, or metabolism.

This study requires a one time 8.5 ml blood sample and clinical data to be obtained at initiation of therapy, 4 months after initiation of therapy and 12 months after initiation of therapy.

DETAILED DESCRIPTION:
This study will make use of a large population of well defined patients with Pulmonary Arterial Hypertension who were enrolled in Encysive Pharmaceutical's STRIDE clinical trials or who have received bosentan or ambrisentan for 4 months or longer. This international study constitutes the largest clinical study of this deadly disease and in such has great potential to alter the clinical practice by revealing novel gene-drug interactions. This study tests the hypothesis by executing the following aims:

Aim 1: Determine in Pulmonary Arterial Hypertension (the relationship between known disease-specific polymorphisms (Serotonin transporter gene and PAI HindIII) and variants in BMPR2 and SMAD4 with several well-defined clinical efficacy endpoints of sitaxsentan, bosentan, and ambrisentan therapy.

Aim 2: Determine in Pulmonary Arterial Hypertension the relationship between existing potentially "therapy-specific" polymorphisms in the ET-1, ETAR, ETBR, NPR-C, prostacyclin receptor and prostacyclin synthase with several well-defined clinical efficacy endpoints of sitaxsentan, bosentan, and ambrisentan therapy.

Aim 3: Characterize the relationship between any treatment effect, these polymorphisms and PAH severity, using either clinical data or clinical surrogates for disease activity.

***This study was funded by the NIH from 2005 - 2009. In August 2009 a no-cost extension was granted and this study continued until the end of July 2010. Currently the study is still active and does still have several active sites participating; however, the study is funded by the internal institution and there is no contributing federal funding.***

ELIGIBILITY:
Inclusion Criteria:

GROUP 1

* Patients have to be currently enrolled or previously enrolled in STRIDE FPH01, FPH01-XC FPH02, FPH02x, FPH03, FPH04 or FPH06.
* WHO Group 1 Pulmonary Arterial Hypertension: Idiopathic, Familial, Associated with (APAH) Collagen vascular disease, congenital systemic-to-pulmonary shunts, portal hypertension, Drugs and toxins (e.g., anorexigens, rapeseed oil, L-tryptophan, methamphetamine, and cocaine), other (thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders, splenectomy) Associated with significant venous or capillary involvement, Pulmonary veno-occlusive disease, Pulmonary-capillary hemangiomatosis.

GROUP 2

* Patients currently receiving bosentan or ambrisentan OR who have previously received bosentan or ambrisentan for greater than 4 (four) months.
* WHO Group 1 Pulmonary Arterial Hypertension: Idiopathic, Familial, Associated with (APAH), collagen vascular disease, congenital systemic-to-pulmonary shunts, portal hypertension, drugs and toxins (e.g., anorexigens, rapeseed oil, L-tryptophan, methamphetamine, and cocaine), other (thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders, or splenectomy), associated with significant venous or capillary involvement, pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis.

Exclusion Criteria:

GROUP 1

* Not enrolled in the Encysive Pharmaceutical's STRIDE study(sitaxsentan).
* Known infectious disease (HIV, Hepatitis).

GROUP 2

* Never enrolled in the STRIDE study for sitaxsentan patients.
* Not currently or previously on bosentan or ambrisentan.
* Patients who were previously on bosentan or ambrisentan must have been on bosentan or ambrisentan for greater than 4 months.
* Known infectious disease (HIV, Hepatitis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must have been diagnosed with WHO Group 1 Pulmonary Arterial Hypertension: Idiopathic, Familial or Associated with (APAH) Collagen vascular disease, congenital systemic-to-pulmonary shunts, portal hypertension, Drugs and toxins , other (thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders, splenectomy) Associated with significant venous or capillary involvement, Pulmonary veno-occlusive disease, Pulmonary-capillary hemangiomatosis. Patients currently therapy must include sitaxsentan, bosentan, or ambrisentan OR patients must have previously been treated with sitaxsentan, bosentan or ambrisentan for 4 months or longer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 12 months after initiation of drug therapy

SECONDARY OUTCOMES:
Hemodynamics - Right Heart Catheterization | 12 months after intitation of drug therapy
Borg | 12 months after initiation of drug therapy
Functional Class - FC | 12 months after intitation of drug therapy
Toxicities | 12 months after initiation of drug therapy
Time of Clinical Worsening | 12 months after initiation of drug therapy
Decline in WHO Functional Class | 12 months after initiation of drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Benza, MD, Principal Investigator — Allegheny General Hospital/Allegheny-Singer Research Institute of West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Pulmonary Hypertension Association website — http://www.phassociation.org